CLINICAL TRIAL: NCT02567682
Title: A Phase 1, Open-Label Study to Evaluate the Effect of Multiple Doses of GBT440 on the Pharmacokinetics of Probe Substrates for CYP1A2, CYP2C9, CYP2C19, and CYP3A4 in Healthy Subjects
Brief Title: Drug Interaction Study of GBT440 With Caffeine, S-warfarin, Omeprazole, and Midazolam in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Global Blood Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBT440-003
Record Dates: First submitted 2015-09-23; First posted 2015-10-05 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Sickle Cell Disease
Keywords: anemia, sickle cell
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — voxelotor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fixed sequence, 2-periods (Experimental): An open-label, fixed sequence, 2-period drug interaction study Period 1 Treatment A: Single dose of drug cocktail on Day 1 Period 2 Treatment B: GBT440 on Days 1 through 3 and Treatment C: Single dose of drug cocktail on Day 4 and GBT440 on Days 4 through 7
  Interventions: Drug: GBT440

INTERVENTIONS:
Drug: GBT440 — GBT440 capsules followed by Caffeine, S-warfarin+vitamin K, Omeprazole, and Midazolam

SUMMARY:
The purpose of this study to evaluate the effect of concomitant administration of GBT440 on caffeine (a CYP1A2 probe substrate), S warfarin (a CYP2C9 probe substrate), omeprazole (a CYP2C19 probe substrate), and midazolam (a CYP3A4 probe substrate) plasma concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a female of non-childbearing potential or male, who is healthy, nonsmoking, and 18 to 55 years old, inclusive, at screening
* Male subjects agree to use contraception
* Willing and able to give written informed consent

Exclusion Criteria:

* Evidence or history of clinically significant metabolic, allergic, dermatological, hepatic, renal,hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder
* History of hypersensitivity or allergy to drugs, foods, or other substances
* History or presence of abnormal electrocardiogram or hypertension
* History of alcohol abuse, illicit drug use, significant mental illness, physical dependence to any opioid, or any history of drug abuse or addiction within 1 year of screening
* Participated in another clinical trial of an investigational drug within 30 days (or 5 half-lives of the investigational drug, whichever is longer) prior to Screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration(Cmax) for caffeine, S warfarin, omeprazole, and midazolam in plasma | 0 - 168 hours post dose in Period 1 and 0-408 hours post dose in Period 2
Area under the plasma concentration-time curve (AUC) from time 0 to the time of the last quantifiable concentration (AUCt) for caffeine, S warfarin, omeprazole, and midazolam | 0 - 168 hours post dose in Period 1 and 0-408 hours post dose in Period 2
Area under the plasma concentration time curve from time 0 extrapolated to infinity (AUCinf) for caffeine, S warfarin, omeprazole, and midazolam | 0 - 168 hours post dose in Period 1 and 0-408 hours post dose in Period 2

SECONDARY OUTCOMES:
The time that Cmax was observed (tmax) for caffeine, S warfarin, omeprazole, and midazolam in plasma | 0 - 168 hours post dose in Period 1 and 0-408 hours post dose in Period 2
Terminal elimination half-life (t½) for caffeine, S warfarin, omeprazole, and midazolam in plasma | 0 - 168 hours post dose in Period 1 and 0-408 hours post dose in Period 2
Cmax for metabolites of caffeine, warfarin, omeprazole, and midazolam in plasma | 0 - 168 hours post dose in Period 1 and 0-408 hours post dose in Period 2
tmax, for metabolites of caffeine, warfarin, omeprazole, and midazolam in plasma | 0 - 168 hours post dose in Period 1 and 0-408 hours post dose in Period 2
AUCt for metabolites of caffeine, warfarin, omeprazole, and midazolam in plasma | 0 - 168 hours post dose in Period 1 and 0-408 hours post dose in Period 2
AUCinf for metabolites of caffeine, warfarin, omeprazole, and midazolam in plasma | 0 - 168 hours post dose in Period 1 and 0-408 hours post dose in Period 2
t1/2 for metabolites of caffeine, warfarin, omeprazole, and midazolam in plasma | 0 - 168 hours post dose in Period 1 and 0-408 hours post dose in Period 2
Ratio of metabolite to parent Cmax corrected for molecular weight (Cmax M/P) for metabolites of caffeine, warfarin, omeprazole, and midazolam in plasma | 0 - 168 hours post dose in Period 1 and 0-408 hours post dose in Period 2
Ratio of metabolite to parent AUCt corrected for molecular weight (AUCt M/P)for metabolites of caffeine, warfarin, omeprazole, and midazolam in plasma | 0 - 168 hours post dose in Period 1 and 0-408 hours post dose in Period 2
Ratio of metabolite to parent AUCinf corrected for molecular weight (AUCinf M/P) for metabolites of caffeine, warfarin, omeprazole, and midazolam in plasma | 0 - 168 hours post dose in Period 1 and 0-408 hours post dose in Period 2
Cmax for GBT440 in whole blood and plasma | 0 - 168 hours post dose in Period 1 and 0-408 hours post dose in Period 2
tmax for GBT440 in whole blood and plasma | 0 - 168 hours post dose in Period 1 and 0-408 hours post dose in Period 2
AUC from time 0 to 24 hours (AUC0-24) (Days 4 and 7) for GBT440 in whole blood and plasma | 0 - 168 hours post dose in Period 1 and 0-408 hours post dose in Period 2
t1/2 (Day7) for GBT440 in whole blood and plasma | 0 - 168 hours post dose in Period 1 and 0-408 hours post dose in Period 2

OTHER OUTCOMES:
Treatment-emergent adverse events (TEAEs) and serious adverse events | Baseline to Period 2 Day 25
Change in clinical laboratory tests | Baseline to Period 2 Day 25
Change in physical examination findings | Baseline to Period 2 Day 25
Change in vital signs | Baseline to Period 2 Day 25
Change in pulse oximetry findings | Baseline to Period 2 Day 25
Change in electrocardiograms (ECGs) | Baseline to Period 2 Day 25

CONTACTS AND LOCATIONS:
Overall Officials: Carla Washington, PhD, Study Director — Global Blood Therapeutics
Locations (1):
- ICON Early Phase Services, LLC Clinical Research Unit, San Antonio, Texas, United States